CLINICAL TRIAL: NCT06916715
Title: Feasibility and Diagnostic Accuracy of Magnetic Resonance Elastography in Intracranial Space-Occupying Lesions
Brief Title: MR Elastography in Intracranial Lesions: Feasibility & Accuracy
Status: Active, not recruiting | Type: Observational
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Yu Shi, Professor, Shengjing Hospital
Other Study IDs: Shengjing_Brain
Record Dates: First submitted 2025-03-31; First posted 2025-04-08 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Brain Neoplasms
Keywords: Magnetic resonance elastography
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intracranial Neoplastic and Non-Neoplastic Lesions: This group encompasses patients with intracranial neoplastic lesions (including low-grade tumors, WHO 1-2; and high-grade tumors, WHO 3-4) and non-neoplastic lesions. It involves retrospective analysis of magnetic resonance elastography (MRE) data to assess the feasibility and diagnostic accuracy of MRE in identifying and differentiating various intracranial pathologies.

SUMMARY:
Brain tumors, despite their relatively low incidence among cancers, are associated with high morbidity and mortality due to the brain's complexity. Biopsy, the gold standard for tumor grading, is limited by invasiveness, costs, and sampling issues. Conventional MR imaging lacks sensitivity to differentiating tumor grades, while magnetic resonance elastography (MRE) offers non-invasive assessment potential. This retrospective study reviewed MRE data from 512 brain tumor patients (May 2017-December 2024) to evaluate MRE's diagnostic performance, success rate in tumor grading, and clinical reliability, aiming to advance its role in non-invasive brain tumor assessment.

DETAILED DESCRIPTION:
Despite their relatively low incidence among all cancers, brain tumors are associated with substantial morbidity and mortality, attributed to the brain's intricate structure and critical physiological roles. Pathologically categorized into meningioma, pituitary adenoma, glioma, craniopharyngioma, germ cell tumor, chordoma, metastatic tumor, acoustic neuroma, and lymphoma, these neoplasms undergo a complex, multi-stage evolution-encompassing initial cellular alterations, tumorigenesis, progression, and potential metastasis. Their oncogenesis is intricately linked to dysregulated cell differentiation during embryonic development, where lower differentiation grades typically correlate with higher malignancy. Clinically, brain tumors manifest as elevated intracranial pressure, neurological and cognitive deficits, and epileptic seizures.

The curability of brain tumors depends on tumor type, grading, and therapeutic strategies. While benign tumors often achieve complete remission through surgical resection, malignant tumors require sophisticated multimodal therapies. Although biopsy serves as the gold standard for tumor grading, its invasive nature, high cost, potential complications, poor patient tolerance, and susceptibility to sampling bias and interpretive subjectivity limit its applicability for frequent monitoring. In this context, non-invasive imaging modalities-such as magnetic resonance elastography (MRE)-capable of longitudinal assessment of lesioned brain tissue, provide invaluable clinical insights, guiding emerging therapeutic interventions aimed at decelerating or halting progression to terminal brain tumors.

Conventional magnetic resonance (MR) imaging effectively visualizes tumors via morphological changes; however, these traditional techniques demonstrate limited sensitivity to differentiating tumor grades. Emerging evidence highlights MRE's potential in tumor grading and diagnosis. Despite the increasing clinical adoption of brain MRE, its widespread implementation remains restricted. Therefore, rigorous quality control of MRE acquisitions is essential to ensure result reproducibility and reliability, while identifying root causes of suboptimal outcomes.

This retrospective study analyzed MRE findings from 512 patients with brain tumors between May 2017 and December 2024. By evaluating MRE's diagnostic efficacy, success rate in tumor grading, and clinical reliability, the research addresses critical gaps in non-invasive brain tumor assessment, contributing to the advancement of evidence-based neuro-oncological imaging practices.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing intracranial space-occupying lesions resection surgery are eligible for inclusion in the study.

Exclusion Criteria:

* Patients with metallic implants or foreign bodies in their bodies (pacemakers, artificial metallic heart valves, metal joints, metal implants, and those who can not remove dentures, insulin pumps, or contraceptive rings)
* Pregnant women in the first trimester (within three months)
* Patients with severe claustrophobia or anxiety
* Patients with severe fever
* Patients who can not tolerate MRE
* Patients with vascular malformations and aneurysms.
* Patients who do not sign an informed consent

Ages: 8 Years to 83 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This retrospective study enrolled 512 patients diagnosed with intracranial space-occupying lesions who underwent magnetic resonance elastography (MRE) at Shengjing Hospital between May 2017 and December 2024. All participants had available MRE data, met inclusion criteria (scheduled for intracranial space-occupying lesion resection surgery and provided written informed consent), and covered diverse intracranial space-occupying lesions , serving as the cohort for MRE-based space-occupying lesions characteristic analysis.
Sampling Method: Non-Probability Sample
Enrollment: 512 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2025-12-09 (Actual); Study Completion 2026-12-09 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of Magnetic Resonance Elastography (MRE) for Brain Tumor Grading | Data collection period: May 2017-December 2024 (retrospective analysis of existing MRE and clinical data).
  Evaluate diagnostic performance of MRE in differentiating brain tumor grades (e.g., WHO grades), using pathological results as the gold standard. Metrics include sensitivity, specificity, and overall diagnostic accuracy.
Success Rate of Magnetic Resonance Elastography (MRE) in Assessing Intracranial Space-Occupying Lesions | Data analysis period: May 2017-December 2024.
  Determine the successful application rate of MRE in acquiring valid imaging data for intracranial space-occupying lesions, analyzing technical feasibility and influencing factors.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Shi, MD, Principal Investigator — Shengjing Hospital; Anhua Wu, MD, Principal Investigator — Shengjing Hospital; Wen Cheng, MD, Principal Investigator — Shengjing Hospital
Locations (1):
- Shengjing Hospital, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yin M, Glaser KJ, Talwalkar JA, Chen J, Manduca A, Ehman RL. Hepatic MR Elastography: Clinical Performance in a Series of 1377 Consecutive Examinations. Radiology. 2016 Jan;278(1):114-24. doi: 10.1148/radiol.2015142141. Epub 2015 Jul 8. PMID 26162026
- [Background] Louis DN, Perry A, Wesseling P, Brat DJ, Cree IA, Figarella-Branger D, Hawkins C, Ng HK, Pfister SM, Reifenberger G, Soffietti R, von Deimling A, Ellison DW. The 2021 WHO Classification of Tumors of the Central Nervous System: a summary. Neuro Oncol. 2021 Aug 2;23(8):1231-1251. doi: 10.1093/neuonc/noab106. PMID 34185076